CLINICAL TRIAL: NCT07335770
Title: Clinical Utility of CMR for Diagnosis, Treatment Guidance and Prognostication of Cardiac Masses
Brief Title: Cardiac Magnetic Resonance for Diagnosis, Treatment Guidance and Prognosis of Cardiac Masses (CMR)
Status: Enrolling by invitation | Type: Observational
Sponsor: Minjie Lu (Other)
Responsible Party: Sponsor-Investigator, Minjie Lu, MD, PhD, Chinese Academy of Medical Sciences, Fuwai Hospital
Organization: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Other Study IDs: CMR_Cardiac Mass
Record Dates: First submitted 2025-12-27; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Masses
Keywords: cardiovascular magnetic resonance; diagnosis; prognosis prediction
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Neoplastic Cardiac Mass Cohort: Patients with histopathologically confirmed or clinically diagnosed neoplastic cardiac masses, including primary cardiac tumors (benign: myxoma, fibroma, rhabdomyoma; malignant: angiosarcoma, rhabdomyosarcoma) and secondary cardiac metastases (from lung cancer, breast cancer, hematological malignancies, etc.). All patients undergo complete CMR evaluation (conventional sequences + quantitative mapping + FPP + LGE) and long-term follow-up.
  Interventions: Diagnostic Test: CMR-Based Tissue Characterization + Lesion-Specific Clinical Management
- Non-Neoplastic Cardiac Mass Cohort: Patients with confirmed non-neoplastic cardiac masses, including cardiac thrombi (diagnosed by anticoagulation response or histopathology), pericardial cysts, inflammatory pseudotumors, etc. All patients complete CMR examinations and follow-up as required.
  Interventions: Diagnostic Test: CMR-Based Tissue Characterization + Lesion-Specific Clinical Management
- Benign Cardiac Mass Cohort: Patients with histopathologically confirmed benign cardiac masses, including myxoma, fibroma, rhabdomyoma, lipoma, pericardial cyst, etc. All undergo complete CMR evaluation and long-term follow-up.
  Interventions: Diagnostic Test: CMR-Based Malignancy Differentiation + Tumor-Nature-Specific Clinical Management
- Malignant Cardiac Mass Cohort: Patients with confirmed malignant cardiac masses, including primary malignant tumors (angiosarcoma, rhabdomyosarcoma) and secondary cardiac metastases (from lung cancer, breast cancer, hematological malignancies, etc.). All complete CMR examinations and follow-up as required.
  Interventions: Diagnostic Test: CMR-Based Malignancy Differentiation + Tumor-Nature-Specific Clinical Management
- Favorable Prognosis Cohort: Patients with cardiac masses (neoplastic/non-neoplastic) who are alive without lesion recurrence, major adverse cardiac events (thromboembolism, heart failure), or progressive cardiac dysfunction at the 3-year follow-up.
  Interventions: Diagnostic Test: CMR-Based Prognostic Stratification + Outcome-Targeted Follow-Up
- Unfavorable Prognosis Cohort: Patients with cardiac masses (neoplastic/non-neoplastic) who experience all-cause death, lesion recurrence, major adverse cardiac events, or progressive cardiac dysfunction during the 3-year follow-up.
  Interventions: Diagnostic Test: CMR-Based Prognostic Stratification + Outcome-Targeted Follow-Up

INTERVENTIONS:
Diagnostic Test: CMR-Based Tissue Characterization + Lesion-Specific Clinical Management — For the neoplastic cohort: Standardized 3.0T CMR (conventional sequences + quantitative mapping + FPP + LGE) to characterize tumor nature (benign/malignant, primary/metastatic) and guide clinical management (surgical resection, chemotherapy, radiotherapy, or surveillance). For the non-neoplastic cohort: CMR to confirm lesion type (thrombus, cyst, etc.) and guide targeted treatment (anticoagulation, surgical excision, anti-inflammatory therapy, or conservative follow-up). All patients complete 3-year long-term follow-up to assess outcomes.
  Groups: Neoplastic Cardiac Mass Cohort; Non-Neoplastic Cardiac Mass Cohort
Diagnostic Test: CMR-Based Malignancy Differentiation + Tumor-Nature-Specific Clinical Management — For the benign cohort: Standardized 3.0T CMR (conventional sequences + quantitative mapping + FPP + LGE) to confirm benign nature and guide clinical management (curative surgical resection for symptomatic/large lesions or long-term surveillance for asymptomatic small lesions). For the malignant cohort: CMR to assess tumor invasiveness, metastasis, and cardiac function impact, further guiding individualized treatment (radical resection, adjuvant chemotherapy/radiotherapy, palliative therapy, or systemic therapy for primary tumors). All patients complete 3-year long-term follow-up to monitor recurrence and survival outcomes.
  Groups: Benign Cardiac Mass Cohort; Malignant Cardiac Mass Cohort
Diagnostic Test: CMR-Based Prognostic Stratification + Outcome-Targeted Follow-Up — For both cohorts: Baseline standardized 3.0T CMR evaluation (conventional sequences + quantitative mapping + FPP + LGE) to collect potential prognostic indicators (lesion size, infiltration extent, enhancement pattern, T1/T2 values, ECV). During 3-year follow-up, regular assessments (outpatient visits, CMR re-evaluation, telephone follow-up) are conducted to monitor outcomes. The intervention focuses on analyzing the correlation between baseline CMR features and prognostic status (favorable/unfavorable) to validate CMR's predictive value for long-term outcomes.
  Groups: Favorable Prognosis Cohort; Unfavorable Prognosis Cohort

SUMMARY:
The goal of this observational study is to explore the diagnostic accuracy, treatment-guiding value, and prognostic predictive utility of cardiovascular magnetic resonance (CMR) in patients with suspected or confirmed cardiac masses. Cardiac masses include neoplastic (primary tumors, secondary metastases) and non-neoplastic (thrombi, pericardial cysts, inflammatory pseudotumors) lesions-primary tumors are extremely rare (incidence: 0.0017%-0.03%), with 75% benign (myxoma accounting for 40%-50%) and 25% malignant (predominantly angiosarcoma), while secondary metastases are 20-40 times more common. Non-neoplastic masses like thrombi are linked to atrial fibrillation and heart failure, with thromboembolism as a fatal complication. Due to non-specific symptoms (chest pain, dyspnea) and pathological heterogeneity, accurate lesion differentiation and outcome prediction remain clinical challenges.

CMR serves as the "silver standard" for non-invasive assessment of cardiac masses, leveraging superior soft tissue resolution, multi-planar imaging, and multi-parameter tissue characterization (T1/T2 weighted imaging, FPP, LGE, T1/T2 mapping, ECV). Multicenter studies confirm its 98.4% overall diagnostic accuracy and 98.4% benign/malignant differentiation accuracy, with excellent consistency with histopathology (Cohen's Kappa = 0.88). However, existing research is mostly retrospective with small samples, lacking systematic validation of quantitative CMR indicators-gaps this study addresses.

The main questions it aims to answer are:

Does CMR (qualitative + quantitative indicators) accurately differentiate neoplastic/non-neoplastic and benign/malignant cardiac masses (gold standard: histopathology or long-term follow-up)? Can CMR features (size, margin, infiltration, enhancement pattern, T1/T2 values, ECV) guide treatment selection (surgical resection, interventional therapy, medical treatment, conservative follow-up)? Do specific CMR indicators independently predict long-term outcomes (all-cause mortality, recurrence, thromboembolism) in patients with cardiac masses? Participants will include patients who undergo CMR for suspected/confirmed cardiac masses Patients receiving routine CMR as part of clinical care will have their CMR images analyzed, treatment plans recorded, and be followed up for 3 years via outpatient visits, telephone, or electronic medical records (at 1, 3, 6, 12, 24, 36 months) to collect survival status, recurrence, cardiac function changes, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected or confirmed cardiac masses by imaging examinations (e.g., echocardiography, computed tomography).
2. Scheduled for or have completed cardiovascular magnetic resonance (CMR) examination.

Exclusion Criteria:

1. Unable to obtain diagnostic-quality cardiac CMR images (due to uncontrollable claustrophobia, severe motion/arrhythmia artifacts, uncorrectable scanning failures).
2. Unable to determine the nature of the cardiac mass (inaccessible to histopathological examination, unclear diagnosis via comprehensive clinical evaluation).
3. Unable to obtain follow-up information (lost to follow-up, refusal of follow-up, unclear outcome attribution due to severe concurrent diseases).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with cardiac mass experienced CMR scanning
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2008-01-01 (Actual); Primary Completion 2035-11-30 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Nature of the mass | 5 years
  The diagnosis of the nature of tumors was established based on histopathology results when these results were available, or alternatively based on the presence of distant metastasis confirmed during follow-up.
All Because of Death | 5 years
  This endpoint is formally referred to as All-Cause Mortality in clinical research; it denotes the occurrence of death in a study participant from any underlying reason (regardless of whether the cause is related to the study's target disease, intervention, or unrelated comorbidities/incidents) during the predefined observation period.
  The approaches of collection of all-cause mortality data outlined below:
  Study teams conduct scheduled follow-ups (e.g., in-clinic visits, telephone check-ins, or remote patient monitoring) at predefined intervals (every 6 months) to inquire about the participant's survival status. Supplemental Verification via Inpatient Record Systems involves querying the hospital's inpatient electronic health record system if the participant is admitted to a hospital during the follow-up period.